CLINICAL TRIAL: NCT06797986
Title: A Phase I/IIa Clinical Trial to Investigate the Safety, Immunogenicity and Efficacy of BVAC-E6E7 in Subjects with HPV Type 16 And/or 18 Positive Unresectable Recurrent or Metastatic Head
Brief Title: A Phase I/IIa Clinical Trial to Investigate BVAC-E6E7 in Subjects with HPV Positive HNSCC.
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cellid Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VIVACE-001
Record Dates: First submitted 2024-11-20; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma (HNSCC); HPV (human Papillomavirus)-Associated Carcinoma; HPV Positive Oropharyngeal Squamous Cell Carcinoma
Keywords: HNSCC; BVAC-E6E7; HPV Type 16 and/or 18 Positive
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- BVAC-E6E7 (low level) (Experimental): Part A (low level) Test group will receive low dose level (2.5 x 10^7 cells/dose) of BVAC-E6E7 for every 3 weeks, 6 times by IV injection
  Interventions: Biological: BVAC-E6E7 (low level)
- BVAC-E6E7 (high level) (Experimental): Part A (high level) Test group will receive high dose level (5.0 x 10^7 cells/dose) of BVAC-E6E7 for every 3 weeks, 6 times by IV injection
  Interventions: Biological: BVAC-E6E7 (high level)
- BVAC-E6E7 (RP2D) (Experimental): Part B Test group will receive RP2D of BVAC-E6E7 for every 3 weeks, 6 times by IV injection
  Interventions: Biological: BVAC-E6E7 (RP2D)

INTERVENTIONS:
Biological: BVAC-E6E7 (low level) — BVAC-E6E7 is an immunotherapeutic vaccine designed to treat unresectable recurrent or metastatic head and neck squamous cell carcinoma positive to HPV 16 or 18.
  Arms: BVAC-E6E7 (low level)
Biological: BVAC-E6E7 (high level) — BVAC-E6E7 is an immunotherapeutic vaccine designed to treat unresectable recurrent or metastatic head and neck squamous cell carcinoma positive to HPV 16 or 18.
  Arms: BVAC-E6E7 (high level)
Biological: BVAC-E6E7 (RP2D) — BVAC-E6E7 is an immunotherapeutic vaccine designed to treat unresectable recurrent or metastatic head and neck squamous cell carcinoma positive to HPV 16 or 18.
  Arms: BVAC-E6E7 (RP2D)

SUMMARY:
BVAC-E6E7 is an immunotherapeutic vaccine designed to treat unresectable recurrent or metastatic head and neck squamous cell carcinoma positive to HPV 16 or 18. This clinical trial for BVAC-E6E7 consists of two phases: PhaseⅠfocuses on safety and tolerance to determine the maximum tolerated dose (MTD), while Phase Ⅱ evaluates its efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male and female aged 19 and above at the time of acquisition informed consent form.
2. Patients who have agreed to provide blood and tissue samples during the clinical trial.
3. Patients with Head and neck squamous cell carcinoma histologically confirmed as HPV type 16 or 18 positive * The biopsy results obtained during screening process or the genotyping (PCR, microarray test) results from stored tissue (formalin-fixed paraffin-embedded) prior to screening should be confirmed positive to HPV type 16 or 18.
4. Patients who are histologically or cytologically diagnosed with recurrent/metastatic Head and neck squamous cell carcinoma (excluding Nasopharyngeal carcinoma).
5. Patients with at least one measurable or evaluable lesion confirmed by CT or MRI according to RECIST v1.1. [It can be considered as an evaluable lesion if the disease has progressed in the previously irradiated area.]
6. Patients who meet one of the following criteria and have no available standard treatment due to contraindication, intolerance or refusal of administration.

   ① Patients who have progressed or recurred the cancer during or after the completion of primary or subsequent platinum based palliative systemic chemotherapy to treat the recurrent or metastatic Head and neck cancer.

   ② Patients who have confirmed the progression of cancer within 24 weeks after the final administration of immune checkpoint blocker (ICI) or completion of combination treatment including platinum agents with a radical purpose.

   ③ Patients who are ineligible for platinum based chemotherapy due to contraindications, intolerance or refusal of administration of platinum based chemotherapy.
7. Patients with ECOG performance status of 0 or 1
8. Patients with at least a 3-month life expectancy.
9. Male patients who has not received the vasectomy should agree usage barrier contraceptive method (i.e. condom) and agree to use appropriate contraception for themselves and their partners for at least 6 months after the completion of IP administration.

   * Appropriate contraceptive method: absolute abstinence, hormone contraceptive agent with unknown drug-interaction (e.g. levonorgestrel intrauterine system (IUS) (Mirena) or Medroxyprogesterone) and surgical sterilization operation (Vasectomy, Bilateral salpingectomy and ligation, etc.). However, Intermittent abstinences (ovulation period, symptothermal method or late-ovulation) or Coitus interruptus are not considered as appropriate contraceptive method.

Exclusion Criteria:

1. Patients with a history of malignant tumor, excluding Head and neck squamous cell carcinoma, within 3 years prior to the screening (However, patients who are judged by investigator to have been cured of Basal cell carcinoma (BCC) / Squamous cell carcinoma (SCC) of the skin, localized prostate cancer, papillary thyroid cancer, or cervical intraepithelial neoplasia (CIN) are able to enroll.)
2. Nasopharyngeal cancer or Head and neck cancer other than squamous cell carcinoma.
3. Patients having below cardiovascular disease at the time of the screening process.

   ① Myocardial infarction or Unstable angina within 6 months prior to the first IP administration (baseline).
   * Severe heart failure or congestive heart failure of class Ⅲ or higher according to the New York Heart Association (NYHA).

     * Ventricular arrhythmia requiring treatment. ④ Severe conduction disorder (e.g. 3rd degree AV block) ⑤ Uncontrolled hypertension according to the judgement by investigator.
4. Patients who have confirmed clinically significant symptoms or uncontrolled central nervous system, brain metastasis, or carcinomatous meningitis (However, patients who have not confirmed the progression disease for at least 4 weeks after central nervous system or metastatic brain treatment and have not required treatment using steroid or other meditation within 7 days prior to the IP administration can be enrolled.)
5. Patients with a history or confirmed active immune disease (e.g. rheumatoid arthritis, inflammatory bowel disease, systemic lupus erythematosus, vasculitis, multiple sclerosis, or T cell lymphoma) after receiving systemic treatment (e.g. disease-modifying agent, corticosteroid or immunosuppressive drug) [However, alternative treatment (thyroxine, insulin, physiologic corticosteroid alternative treatment due to dysfunction of adrenal gland or pituitary gland) are not considered as systemic treatments.]
6. Patients who are unable to collect the blood for production of the IP, according to the judgement of investigator, due to thromboembolism disease or bleeding diatheses.
7. Patients with a positive human immunodeficiency virus (HIV) test result
8. Patients with active hepatitis B or C according to the hepatitis B virus (HBV) and hepatitis C virus (HCV) test result.

   ① Patients positive for HBsAg and HBV DNA.

   ② Patients positive for anti-HCV and HCV RNA.
9. Patients with autoimmune disease or history of chronic or recurrent autoimmune diseases.
10. Patients with a history of organ transplantation.
11. Hematopoietic stem cell transplantation (HSCT) patients.
12. Patients who have confirmed severe or uncontrolled active inflammation within 12 weeks prior to screening process.
13. Patients with a history of hypersensitivity to the components of IP.
14. Patients who have administrated a leukocyte product within 12 weeks prior to screening process.
15. Patients who have received chemotherapy, radiotherapy or targeted therapy within 4 weeks prior to baseline [However, patients who have not recovered to NCI-CTCAE v5.0 Grade 1 or baseline levels from chemotherapy-related toxicities. (excluding Alopecia and vitiligo), even after 4 weeks, are not eligible for enrollment.]
16. Patients who have administrated live-vaccine or live attenuated vaccine within 4 weeks prior to baseline.
17. Patients who have administrated immunosuppressant within 2 weeks prior to baseline. (However, usage corresponding to the following immunosuppressant is allowed.)

    * Steroid for nasal cavity, aspiration, topical, or local site (e.g. Intra-articular injection)
    * Prednisolone 10 mg/day or systemic corticosteroid at a physiologic dose that does not exceed the equivalent amount.
    * Steroids used for pretreatment of hypersensitivity (e.g. pretreatment of CT)
18. Patients who meet the following laboratory test standards in the screening test

    * ANC < 1,500/mm³
    * Platelet count < 75,000/mm³
    * Hemoglobin < 9.0 g/dL (If the hemoglobin recovers above 9.0g/dL during the screening period, the patient is eligible for enrollment. However, blood transfusions within 7 days before screening to meet that standard is not allowed.)
    * Serum creatinine >1.5 × ULN
    * Total bilirubin >1.5 × ULN
    * AST or ALT >2.5 × ULN (If liver metastasis confirmed >5 × ULN)
19. Pregnant or lactating women
20. Patients who have administrated IP for other clinical trials or applied investigational device within 4 weeks before screening. [However, the patients who correspond to one of the following, even after 4 weeks, are not eligible for enrollment.]

    ① Patients who have participated in a clinical trial of immune therapeutic vaccine within 1 year before the screening or in an immunotherapy clinical trial within 6 weeks before the screening.

    ② Patients with adverse drug reaction of Grade 2 or higher clearly associated with a previously participated immunotherapy clinical trial.
21. Patients who are not eligible to enroll in this clinical trial according to the judgement of investigator for any other reason.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
[Part A] Incidence of dose-limiting toxicity (DLT) after BVAC-E6E7 administration | On day 1 of cycle 3 (each cycle is 21 days)
  The DLT assessment criteria are based on NCI-CTCAE v5.0. The assessment includes individual criteria for hematologic/non-hematologic toxicities and other toxicities.
  DLT (dose-limiting toxicity) is defined as adverse events or abnormal laboratory values that limit the IP's dose-escalation and are not related to disease progression or intercurrent disease.
[Part B] Objective Response Rate (ORR) | During entire clinical trial, an average of 18 months.
  The ratio of subjects assessed with complete response (CR) or partial response (PR) as a best overall response.
[Part B] Disease Control Rate (DCR) | During entire clinical trial, an average of 18 months.
  The ratio of subjects assessed with CR or PR or stable disease (SD) as a best overall response.
[Part B] Duration of Response (DOR) | From the date of objective response (CR or PR) to the date of disease progression or death, assessed up to 18 months.
  Duration from objective response (CR or PR) to disease progression or death in subjects assessed with CR or PR as a best overall response.
[Part B] 6-month Progression Free Survival rate (PFS rate) or PFS | 6-month after the first IP administration for 6-month PFS / From first IP administration to disease progression or death for PFS
  6-month PFS rate is defined as the ratio of subjects assessed with no disease progression or death at 6 months after the first IP administration.
  PFS is defined as the duration until disease progression or death in subjects from the first IP administration.
[Part B] 12-month Overall Survival rate (OS rate) or OS | 12-month after the first IP administration for 12-month OS rate / From first IP administration to death for OS
  12-month OS rate is defined as the survival rate at 12-month after the first IP administration.
  OS is defined as the duration until death in subjects from the first IP administration.

SECONDARY OUTCOMES:
[Part A] Objective Response Rate (ORR) | During entire clinical trial, an average of 18 months.
  The ratio of subjects assessed with complete response (CR) or partial response (PR) as a best overall response.
[Part A] Disease Control Rate (DCR) | During entire clinical trial, an average of 18 months.
  The ratio of subjects assessed with CR or PR or stable disease (SD) as a best overall response.
[Part A] Duration of Response (DOR) | From objective response (CR or PR) to disease progression or death, assessed up to 18 months.
  Duration from objective response (CR or PR) to disease progression or death in subjects assessed with CR or PR as a best overall response.
[Part A] 6-month Progression Free Survival rate (PFS rate) or PFS | 6-month after the first IP administration for 6-month PFS rate / From first IP administration to disease progression or death for PFS
  6-month PFS rate is defined as the ratio of subjects assessed with disease progression or death at 6 months after the first IP administration.
  PFS is defined as the duration until disease progression or death in subjects from the first IP administration.
[Part A] 12-month Overall Survival rate (OS rate) or OS | 12-month after the first IP administration for 12-month OS rate / From first IP administration to death for OS
  12-month OS rate is defined as the survival rate at 12-month after the first IP administration.
  OS is defined as the duration until death in subjects from the first IP administration.
[Part A/B] Adverse event | During entire clinical trial, an average of 18 months.
  Every adverse event collected from the entire clinical trial is categorized by severity, causality, treatment, or outcome of each adverse event.
[Part A/B] A number of subjects demonstrating abnormal CS in clinical laboratory test | At screening visit, day 1 of every cycle, day 2 of cycle 6 (each cycle is 21 days).
  Clinical laboratory test including hematology, blood chemistry, urinalysis, virus test (only at screening visit).
[Part A/B] A number of subjects demonstrating abnormal CS in vital sign | At screening visit and every visit from the first IP administration day, assessed up to 18 months.
  Vital sign including measure blood pressure, pulse rate, and body temperature
[Part A/B] A number of subjects demonstrating abnormal CS in physical examination | At screening visit, day 1 of cycle 1, Day 2 of Cycle 6 (each cycle is 21 days). If necessary, it can be conducted according to judgement of investigator at other visits from the first IP administration day, assessed up to 18 months.
  The physical examination including examination of the appearance, skin, head/neck, chest/lungs, heart, abdomen, genitourinary/reproductive system, extremities, musculoskeletal system, nervous system, lymph nodes, and other organ.
[Part A/B] A number of subjects demonstrating abnormal CS in 12-lead ECG | At screening visit, day 2 of cycle 6 (1 cycle is 21 days). If necessary, it can be conducted at other visits after first IP administration day until day 1 of cycle 6.
[Part A/B] Detection of E6E7 recombinant gene | At screening visit, day 1 of cycle 1 and day 2 of every cycle (each cycle is 21 days).
  Assesses whether the E6E7 recombinant gene is detected in peripheral blood by BVAC-E6E7 monitoring
[Part A/B] T cell response | At day 1 of cycle 1, day 2 of every cycle, and week 24, 42, 60 after first IP administration (each cycle is 21 days).
  Spot Forming Units (SFU) counts
[Part A/B] Cytokines in the blood | At day 1 of cycle 1, day 2 of every cycle (each cycle is 21 days).
  Concentration changes of IFN-γ, TNF-α, IL-4
[Part A/B] Concentration changes of tumor infiltrating lymphocyte (TIL) in lesion | (optional) at screening visit, day 2 of cycle 6 (each cycle is 21 days).

IPD SHARING:
Plan to Share IPD: Undecided